CLINICAL TRIAL: NCT02510599
Title: An Open Label, Proof of Principle Study to Evaluate the Efficacy and Safety of Solithromycin for the Treatment of Nonalcoholic Steatohepatitis Without Cirrhosis
Brief Title: Safety and Efficacy of Solithromycin in the Treatment of Nonalcoholic Steatohepatitis Without Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE01-205
Record Dates: First submitted 2015-07-01; First posted 2015-07-29 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: NASH; Liver disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases | interventions — solithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Solithromycin (Experimental): Solithromycin 200 mg PO QD for 1 week, followed by 200 mg PO TIW for 12 weeks
  Interventions: Drug: solithromycin

INTERVENTIONS:
Drug: solithromycin
  Other Names: CEM-101

SUMMARY:
The purpose of this study is to evaluate the effects of solithromycin on hepatic histology and biomarkers in patients with nonalcoholic steatohepatitis.

DETAILED DESCRIPTION:
Patients will be administered solithromycin for 13 weeks with regular safety visits and liver biopsies at baseline and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologic evidence of NASH based on liver biopsy obtained within 180 days
* NAS> or = 5
* Able to swallow capsules intact

Exclusion Criteria:

* Symptoms of acute liver disease
* Cirrhosis on liver biopsy
* Positive HIV or Hepatitis tests
* Primary Biliary Cirrhosis
* Poorly controlled diabetes with HgA1C >8.5%
* ALT >4-fold upper limit of normal
* QTcF >450 msec
* CrCl <40 mL/min

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
To evaluate effects on hepatic histology in patients with NASH | 13 weeks
  Using the Nonalcoholic fatty liver disease (NAFLD) Activity Score (NAS)

SECONDARY OUTCOMES:
Changes in Steatosis on liver biopsy | 13 weeks
  Graded from 0 to 3
Changes in hepatocellular ballooning score on liver biopsy | 13 weeks
  Graded from 0 to 2
Changes in inflammation on liver biopsy | 13 weeks
  Graded from 0 to 3

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dobbins, MD, PhD, Study Director — Melinta Therapeutics, Inc.
Locations (1):
- Case Western University Hospitals, Cleveland, Ohio, United States